CLINICAL TRIAL: NCT06917339
Title: Retrospective Analyses Evaluating the Real-World Effectiveness of NeuroStar® TMS and the Factors Associated With Clinical Outcomes
Brief Title: Retrospective Analyses of TrakStar Database
Status: Recruiting | Type: Observational
Sponsor: Neuronetics (Other)
Responsible Party: Sponsor
Other Study IDs: 11-10000-000
Record Dates: First submitted 2025-03-18; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Depression; Obsessive-Compulsive Disorder; Anxiety Depression
Keywords: TMS
MeSH Terms: conditions — Depression; Obsessive-Compulsive Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients treated with NeuroStar TMS
  Interventions: Device: NeuroStar Advanced TMS Therapy System

INTERVENTIONS:
Device: NeuroStar Advanced TMS Therapy System — non-invasive brain stimulation device

SUMMARY:
In this study, real-world data will be used to better understand the effects patient characteristics, symptoms and TMS protocol parameters have on clinical outcomes with NeuroStar TMS.

ELIGIBILITY:
Inclusion Criteria:

* Male or female reported in database and not an invalid entry
* Age reported and not an invalid entry
* Treatment date of November 01, 2008 or later.

Exclusion Criteria:

• Incomplete information on treatment parameters

Ages: 5 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients treated with NeuroStar Advanced TMS Therapy on or after November 1, 2008, and whose treatment information was entered in the Neuronetics TrakStar database.
Sampling Method: Probability Sample
Enrollment: 156000 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2035-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Change in clinical assessment score from baseline to post-treatment | 8 weeks
  real-world efficacy of NeuroStar TMS in reducing patients' symptoms, reduction in clinical assessment score like PHQ-9

SECONDARY OUTCOMES:
Age at baseline and its correlation to change in score post treatment | 8 weeks
  Determine the patient characteristics like age that are associated with clinical outcomes- PHQ-9 following NeuroStar TMS

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor Cole, PhD, Study Director — Neuronetics
Locations (1):
- Neuronetics, Malvern, Pennsylvania, United States